CLINICAL TRIAL: NCT03128489
Title: Immunogenicity and Safety of GSK Biologicals' DTPa-IPV/Hib Conjugate Vaccine (Infanrix™-IPV/Hib) (SB213503) in Healthy Indian Infants
Brief Title: Evaluation of Immunogenicity and Safety of DTPa-IPV/Hib Conjugate Vaccine (Infanrix™-IPV/Hib) Administered at 6, 10 and 14 Weeks in Healthy Indian Infants
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is cancelled due to reassessment of the medical need for the vaccine in India. Cancellation is not related to vaccine's safety and/or efficacy.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201124; 2013-004361-14 (EudraCT Number)
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Diphtheria; Acellular Pertussis; Haemophilus Influenzae Type b; Tetanus; Poliomyelitis
Keywords: Safety; Infanrix™-IPV/Hib; Immunogenicity; Indian infants; Combined vaccine
MeSH Terms: conditions — Diphtheria; Haemophilus Infections; Tetanus; Poliomyelitis | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DTPa-IPV/Hib Group (Experimental): All subjects will receive three doses of primary vaccination at 6, 10 and 14 weeks of age.
  Interventions: Biological: Infanrix-IPV/Hib

INTERVENTIONS:
Biological: Infanrix-IPV/Hib — Subjects will receive (Infanrix-IPV/Hib) as three-dose primary vaccination course at 6, 10 and 14 weeks of age. The vaccine will be administered intramuscularly, at a 90-degree angle into the anterolateral side of the thigh on the right side. The vaccine should not be administered in the buttock.

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of DTPa-IPV/Hib when administered at 6, 10 and 14 weeks to healthy Indian infants, as per guidance from the Indian regulatory authority. The 6, 10 and 14 week schedule reflects the current Indian standard of care.

DETAILED DESCRIPTION:
* Experimental design: Phase III, open-label, non-randomised, multi-centric, single-country study with a single group.
* Duration of the study: The intended duration of the study will be approximately 3 months per subject.
* Treatment group and vaccination schedule: All subjects will receive three doses of the vaccine at 6, 10 and 14 weeks of age.

  * DTPa-IPV/Hib Group: Subjects who will receive DTPa-IPV/Hib vaccine (Infanrix-IPV/Hib).

Other routine registered childhood vaccinations as part of National Immunisation Programme are permitted. Information regarding vaccine administered since birth until study completion will be collected and documented.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representatives [LARs] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 9 weeks of age (42-69 days) at the time of the first vaccination.
* Written informed consent obtained from the parents/LARs of the subject prior to performing any study specific procedure.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born full-term [i.e., after a gestation period of 37 to less than 42 completed weeks (259 to 293 days)].

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before first dose of study vaccine (Day-29 to Day 0), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs from birth to within six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone (0.5 mg/kg/day, or equivalent). Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and 30 days after the last dose of vaccine with the exception of human rotavirus vaccine, hepatitis B vaccine, pneumococcal conjugate vaccine and other vaccines given as a part of the national immunisation schedule, that are allowed at any time during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* History of diphtheria, tetanus, pertussis, poliomyelitis and Hib disease.
* Evidence of previous diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Hib vaccination or disease prior to study enrolment, with the exception of a birth dose of hepatitis B and/or Baccillus Calmette-Guerin (BCG) vaccines and/or oral poliovirus (OPV) vaccine as per local standard of care. The BCG vaccination should occur at least 30 days prior to first dose of vaccination in the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥37.5°C/99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C/100.4°F for rectal route.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of seroprotected subjects in terms of anti-diphtheria (anti-D) and anti-tetanus (anti-T) antibodies. | One month after the third dose of primary vaccination (Month 3)
  A seroprotected subject is a subject whose anti-D/anti-T antibody concentration is greater than or equal to (≥) 0.1 International Units per millilitre (IU/ml).
Number of seroprotected subjects in terms of anti-poliomyelitis (anti-Polio) types 1, 2 and 3 antibodies. | One month after the third dose of primary vaccination (Month 3)
  A seroprotected subject is a subject whose anti-Polio 1, 2 and 3 antibody titers are greater than or equal to (≥) 8 median effective dose (ED50).
Number of seroprotected subjects in terms of anti-polysaccharide Polyribosyl-Ribitol Phosphate (anti-PRP) antibodies. | One month after the third dose of primary vaccination (Month 3)
  A seroprotected subject is a subject whose anti-PRP antibody concentration is greater than or equal to (≥) 0.15 micrograms per millilitre (µg/ml).
Number of subjects with vaccine response to pertussis toxoid (PT), Filamentous Haemagglutinin (FHA) and pertactin (PRN) antigens. | One month after the third dose of primary vaccination (Month 3)
  Vaccine response to pertussis antigens is defined as the appearance of antibodies in subjects who were initially seronegative (i.e., with concentrations lesser than the assay cut-off value), or maintenance of pre-vaccination antibody concentrations in subjects who were initially seropositive (i.e., with concentrations ≥ assay cut-off value).

SECONDARY OUTCOMES:
Anti-D and anti-T antibody concentrations. | One month after the third dose of primary vaccination (Month 3).
  Antibody concentrations are expressed as geometric mean concentrations (GMCs).
Anti-Polio type 1, 2 and 3 antibody titres. | One month after the third dose of primary vaccination (Month 3)
  Antibody titres are expressed as geometric mean titres (GMTs).
Anti-PRP antibody concentrations. | One month after the third dose of primary vaccination (Month 3).
  Antibody concentrations are expressed as geometric mean concentrations (GMCs).
Anti-PT, anti-FHA and anti-PRN antibody concentrations. | One month after the third dose of primary vaccination (Month 3)
  Antibody concentrations are expressed as geometric mean concentrations (GMCs).
Number of seropositive subjects in terms of anti-PT, anti-FHA and anti-PRN antibodies. | One month after the third dose of primary vaccination (Month 3).
  A seropositive subject is a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations above the cut-off value of 5 Enzyme-linked immunosorbent assay (ELISA) Units per millilitre (EL.U/mL).
Anti-PT, anti-FHA and anti-PRN antibody concentrations. | Before the first dose of primary vaccination (Day 0)
  Antibody concentrations are expressed as geometric mean concentrations (GMCs).
Anti-Polio type 1, 2 and 3 antibody titres. | Before the first dose of primary vaccination (Day 0)
  Antibody titres are expressed as geometric mean titres (GMTs).
Anti-PRP antibody concentrations. | Before the first dose of primary vaccination (Day 0)
  Antibody concentrations are expressed as geometric mean concentrations (GMCs).
Number of seropositive subjects in terms of anti-PT, anti-FHA and anti-PRN antibodies. | Before the first dose of primary vaccination (Day 0)
  A seropositive subject is a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations above the cut-off value of 5 EL.U/mL.
Number of seroprotected subjects in terms of anti-Polio type 1, 2 and 3 antibodies. | Before the first dose of primary vaccination (Day 0)
  A seroprotected subject is a subject whose anti-Polio 1, 2 and 3 antibody titers are greater than or equal to (≥) 8 ED50.
Number of seroprotected subjects in terms of anti-PRP antibodies. | Before the first dose of primary vaccination (Day 0)
  A seroprotected subject is a subject whose anti-PRP antibody concentration is greater than or equal to (≥) 0.15 µg/ml.
Number of subjects with solicited local symptoms. | During the 4-day period (Days 0-3) following each vaccination.
  Solicited local symptoms assessed are pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevents normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimetres (mm) of injection site.
Number of subjects with solicited general symptoms. | During the 4-day period (Days 0-3) following each vaccination.
  Solicited general symptoms assessed are drowsiness, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], irritability/fussiness and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevents normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Number of subjects with unsolicited adverse events (AEs). | During the 31-day period (Days 0-30) following each vaccination.
  An unsolicited adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of subjects with serious adverse events (SAEs). | From dose 1 (Day 0) until study end (Month 3)
  Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.